CLINICAL TRIAL: NCT00141219
Title: A 10-Week, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Pregabalin (150 mg - 600 mg/Day) Using a Flexible, Optimized Dose Schedule in Subjects With Peripheral Neuropathic Pain
Brief Title: Pregabalin Peripheral Neuropathic Pain Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081037
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2009-03-13 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2009-09

CONDITIONS: Diabetic Neuropathies; Neuralgia
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: pregabalin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin — 150-600mg/day, BID
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
To evaluate the efficacy of pregabalin, using a flexible, optimized dose schedule with dose adjustment based on Daily Pain Rating Scale (DPRS), compared to placebo in subjects with peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peripheral neuropathic pain syndrome, including diabetic peripheral neuropathy (DPN), postherpetic neuralgia (PHN), or post-traumatic neuropathic pain (including post-surgical), confirmed by a qualified pain specialist.
* Subjects must have completed at least 4 daily pain diaries during the 7 days prior to Visit 2 and have an average pain score of ≥4 over the 7 days prior to Visit 2 (randomization).

Exclusion Criteria:

* Neurologic disorders unrelated to DPN, PHN, or post-traumatic neuropathic pain (including post-surgical), that may confuse or confound the assessment of neuropathic pain.
* Presence of any severe pain associated with conditions other than DPN, PHN, or post-traumatic neuropathic pain (including post-surgical) that may confound the assessment or self evaluation of the pain due to DPN, PHN, or post-traumatic neuropathic pain (including post-surgical).
* Creatinine clearance < 30 mL/min (estimated from serum creatinine, body weight, age, and sex using the Cockcroft and Gault equation in Appendix E). Maximum dose for subjects with creatinine clearance of 30 to 60 mL/min is 300 mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- South Korea (6):
  - Pfizer Investigational Site, Sungnam-si, Gyeonggi-do
  - Pfizer Investigational Site, Suwon, Gyeonggi-do
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081037&StudyName=Pregabalin%20Peripheral%20Neuropathic%20Pain%20Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation and Completion Dates: 27 December 2005 to 28 December 2007; 10 study centers in Korea
Pre-assignment Details: 241 subjects were assigned to study treatment; one subject was randomized but did not receive any study treatment with the reason 'Did not meet entrance criteria'.
Groups:
- Pregabalin: Dose levels of pregabalin were 150 mg/day, 300 mg/day, 450 mg/day, and 600 mg/day which were achieved by taking 75 mg, 150 mg, 225 mg (which was the combination of 75 mg + 150 mg) or 300 mg of pregabalin twice daily (BID), with or without food, once in the morning and once in the evening.
- Placebo: Subjects who were randomized to placebo remained on placebo throughout the remainder of the study.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 162 | 78
Completed | 138 | 62
Not Completed | 24 | 16
Not completed — Protocol violations | 5 | 4
Not completed — Adverse Event | 8 | 6
Not completed — Lack of Efficacy | 5 | 4
Not completed — Withdrawal by Subject | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 162 | 78 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (10.8) | 61.3 (12.9) | 60.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 46 | 129
  Male | 79 | 32 | 111

OUTCOME MEASURES:

1. Secondary Outcome: Daily Pain Rating Scale (DPRS)- Number of 30% Responders (With Respect to Pain Scores)
Description: DPRS consists of an 11-point rating scale ranging from 0 (no pain) to 10 (worst possible pain). A 30% responder at endpoint is a subject who has a 30% or more reduction in mean pain score at endpoint compared to baseline
Time Frame: Endpoint- Week 8 or Early Discontinuation
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. For subjects who did not complete the study, the last 7 available daily pain scores while on study medication were carried forward (LOCF) to calculate the endpoint mean score.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 161 | 77
participants
  Yes | 68 | 27
  No | 93 | 50
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis of no treatment difference in each of the centers; Test type: Superiority or Other; p = 0.289, Cochran-Mantel-Haenszel — All statistical testing was 2-sided and was conducted at the 5% level of significance; P-value in above table was from Cochran-Mantel-Haenszel test comparing Pregabalin and Placebo adjusted for center; Risk Ratio (RR) = 1.115, 95% CI [0.785 to 1.583] — RR estimates relative responder rate between Pregabalin and Placebo (the ratio of the former responder rate to the latter). Estimated RR was center-adjusted ie, assumed common RR in all centers, then a weighted average of center specific RRs computed

2. Secondary Outcome: Daily Pain Rating Scale (DPRS)- Number of 50% Responders (With Respect to Pain Scores)
Description: DPRS consists of an 11-point rating scale ranging from 0 (no pain) to 10 (worst possible pain). A 50% responder at endpoint is a subject who has a 50% or more reduction in mean pain score at endpoint compared to baseline.
Time Frame: Endpoint- Week 8 or Early Discontination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 161 | 77
participants
  Yes | 42 | 11
  No | 119 | 66
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis of no treatment difference in each of the centers; Test type: Superiority or Other; p = 0.041, Cochran-Mantel-Haenszel — All statistical testing was 2-sided and was conducted at the 5% level of significance; P-value in above table was from Cochran-Mantel-Haenszel test comparing Pregabalin and Placebo adjusted for center; Risk Ratio (RR) = 1.644, 95% CI [0.915 to 2.954] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Daily Pain Rating Scale (DPRS)- Mean Pain Score (ITT Population)
Description: DPRS is 11-point rating scale from 0 (no pain) to 10 (worst possible pain). Subjects instructed to describe their pain (daily upon awakening) during preceding 24 hrs by choosing the appropriate number between 0-10. Mean endpoint pain score was obtained from the last 7 available DPRS scores of the daily pain diary while subject on study medication.
Time Frame: Endpoint- Week 8 or Early Discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 161 | 77
score on scale | 4.63 (0.15) [4.33 to 4.92] | 5.13 (0.21) [4.71 to 5.54]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypotheses stated there was no difference in pregabalin and placebo in the primary endpoint versus the alternative that there was. The target sample size was 234 subjects (156 and 78 respectively pregabalin vs placebo using a 2:1 ratio). The calculations assumed a 2-sided comparison at 0.05 alpha, 80% power and 3% dropout. Also, a treatment difference of 1 point and a standard deviation for endpoint mean pain scores of 2.5 were assumed based on previous studies; Test type: Superiority or Other; p = 0.049, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from the general linear model with treatment and center fitted as factors and the baseline value as a covariate; Mean Difference (Final Values) = -0.50, 95% CI [-1.00 to -0.00], Standard Error of Mean 0.252
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; This was a supportive analysis of the primary endpoint to determine if the main results were generalizable across centers; Test type: Superiority or Other; p = 0.729, General Linear Model — Interaction p-value based on adding interaction term to the main model; In supportive model 1, a "treatment by center" independent variable added to the main model
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; This was a supportive analysis of the primary endpoint to determine if the main results were generalizable across different baseline values; Test type: Superiority or Other; p = 0.979, General Linear Model — Interaction p-value based on adding interaction term to the main model; In supportive model 2, a "treatment by baseline mean pain" independent variable added to the main model

4. Other Pre Specified Outcome: Daily Pain Rating Scale (DPRS)- Mean Pain Scores (Evaluable Population)
Description: as for outcome 3
Time Frame: Endpoint- Week 8 or Early Discontinuation
Population: Evaluable (EVAL) Population: Subset of ITT subjects with ≥4 daily pain diaries in the 7 days before Visit 2 (randomization) with average score ≥4; ≥14 days of treatment; ≥14 days of DB daily pain diaries; not withdrawn due to "Protocol violation" or "Did not meet entrance criteria"; not previously participated in the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 149 | 68
score on scale | 4.47 (0.156) [4.16 to 4.78] | 4.94 (0.225) [4.50 to 5.39]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Endpoint Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.077, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center fitted as factors and the baseline value as a covariate; Mean Difference (Final Values) = -0.48, 95% CI [-1.00 to 0.05], Standard Error of Mean 0.267

5. Secondary Outcome: Daily Pain Rating Scale (DPRS)- Weekly Mean Pain Score
Description: DPRS is 11-point rating scale (0=no pain to 10=worst possible pain). Subjects instructed to describe pain (upon awakening) during preceding 24 hrs by choosing appropriate number between 0-10. Mean endpoint pain score obtained from last 7 available DPRS scores of daily pain diary while subject on study medication. Overall Comparison=8-week average.
Time Frame: Weeks 1 to 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. Missing Weekly mean scores were not imputed. Number of subjects analyzed differed by week; noted as n= (pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 162 | 78
score on scale
  Overall Comparison (weeks 1 to 8) | 4.91 (0.110) | 5.29 (0.156)
  Week 1 (n=161, 77) | 5.80 (0.124) | 6.18 (0.176)
  Week 2 (n=156, 75) | 5.30 (0.125) | 5.61 (0.177)
  Week 3 (n=154, 72) | 5.02 (0.125) | 5.42 (0.178)
  Week 4 (n=151, 68) | 4.84 (0.125) | 5.27 (0.180)
  Week 5 (n=146, 66) | 4.69 (0.126) | 5.11 (0.181)
  Week 6 (n=145, 65) | 4.64 (0.126) | 4.93 (0.181)
  Week 7 (n=142, 62) | 4.52 (0.126) | 4.87 (0.183)
  Week 8 (n=138, 62) | 4.47 (0.127) | 4.92 (0.183)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Mean Pain Score Weeks 1 to 8 Overall Comparison (8-week average) Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.042, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from a linear mixed model with treatment, week, center, and treatment by week interaction as factors and baseline value as a covariate; Mean Difference (Final Values) = -0.38, 95% CI [-0.75 to -0.01], Standard Error of Mean 0.186
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 1 Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.071, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from a linear mixed model with treatment, week, center and treatment by week interaction as factors and baseline value as a covariate; Mean Difference (Final Values) = -0.38, 95% CI [-0.79 to 0.03], Standard Error of Mean 0.210
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 2 Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.149, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.31, 95% CI [-0.72 to 0.11], Standard Error of Mean 0.212
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 3 Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.057, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.41, 95% CI [-0.82 to 0.01], Standard Error of Mean 0.213
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 4 Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.044, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.43, 95% CI [-0.85 to -0.01], Standard Error of Mean 0.215
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 5 Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.051, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.42, 95% CI [-0.85 to 0.00], Standard Error of Mean 0.216
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 6 Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.178, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.29, 95% CI [-0.72 to 0.13], Standard Error of Mean 0.216
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 7 Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.104, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.35, 95% CI [-0.78 to 0.07], Standard Error of Mean 0.218
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Week 8 Mean Pain Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.039, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.45, 95% CI [-0.88 to -0.02], Standard Error of Mean 0.218

6. Secondary Outcome: Duration Adjusted Average Change (DAAC) of (Adjusted) Mean Pain Score
Description: DAAC is a score used to assess treatment effects averaged over the entire length of the study. DAAC from baseline to weekly mean pain score was derived by calculating the mean of all post-baseline scores minus baseline mean pain score, and then weighing this according to the proportion of the planned study duration the subject actually completed.
Time Frame: Weeks 1 to 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. Subjects without any post-baseline daily pain scores would have no DAAC; missing DAACs were not imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 161 | 77
score on scale | -1.27 (0.110) [-1.48 to -1.05] | -0.89 (0.156) [-1.20 to -0.58]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Duration Adjusted Average Change (DAAC) Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.044, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = -0.38, 95% CI [-0.74 to -0.01], Standard Error of Mean 0.186

7. Secondary Outcome: Mean Sleep Interference Score Based on Daily Sleep Interference Scale (DSIS).
Description: DSIS consists of an 11-point rating scale (0 = pain did not interfere with sleep to 10 = completely interfered with sleep). Higher score indicating greater level of sleep disturbance.
Time Frame: Endpoint- Week 8 or Early Discontinuation
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. For subjects who did not complete the study, the last 7 available daily sleep interference scores while on study medication were carried forward (LOCF) to calculate the endpoint mean score.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 161 | 77
score on scale | 3.26 (0.162) [2.94 to 3.57] | 3.91 (0.228) [3.46 to 4.36]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Endpoint Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.018, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = -0.65, 95% CI [-1.19 to -0.11], Standard Error of Mean 0.272

8. Secondary Outcome: Mean Sleep Score as Computed by DSIS.
Description: DSIS consists of an 11-point rating scale ranging from 0 = pain did not interfere with sleep to 10 = pain completely interfered with sleep. Overall Comparison= 8-week average.
Time Frame: Weeks 1 to 8
Population: ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. Missing Weekly mean scores were not imputed. Number of subjects analyzed differed by week; noted as n = (pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 162 | 78
score on scale
  Overall Comparison (Weeks 1 to 8) | 3.46 (0.134) | 3.97 (0.189)
  Week 1 (n= 161, 77) | 4.18 (0.145) | 4.56 (0.205)
  Week 2 (n=156, 75) | 3.74 (0.145) | 4.24 (0.206)
  Week 3 (n=154, 72) | 3.55 (0.146) | 4.13 (0.207)
  Week 4 (n=151, 68) | 3.41 (0.146) | 3.95 (0.208)
  Week 5 (n=146, 66) | 3.29 (0.146) | 3.73 (0.209)
  Week 6 (n=145, 65) | 3.22 (0.147) | 3.74 (0.210)
  Week 7 (n=142, 62) | 3.19 (0.147) | 3.71 (0.211)
  Week 8 (n=138, 62) | 3.10 (0.147) | 3.72 (0.211)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Weeks 1 to 8 Mean Sleep Score Overall Comparison (8-week average) Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.024, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.51, 95% CI [-0.96 to -0.07], Standard Error of Mean 0.226
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 1 Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.120, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.38, 95% CI [-0.86 to 0.10], Standard Error of Mean 0.245
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 2 Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.041, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.51, 95% CI [-0.99 to -0.02], Standard Error of Mean 0.246
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 3 Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.017, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.59, 95% CI [-1.07 to -0.10], Standard Error of Mean 0.248
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 4 Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.033, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.53, 95% CI [-1.02 to -0.04], Standard Error of Mean 0.249
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 5 Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.078, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.44, 95% CI [-0.93 to 0.05], Standard Error of Mean 0.250
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 6 Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.038, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.52, 95% CI [-1.01 to -0.03], Standard Error of Mean 0.250
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 7 Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.037, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.53, 95% CI [-1.02 to -0.03], Standard Error of Mean 0.252
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Week 8 Sleep Interference Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.015, Linear Mixed Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; [statistical method as in outcome 5, analysis 2]; Mean Difference (Final Values) = -0.61, 95% CI [-1.11 to -0.12], Standard Error of Mean 0.252

9. Secondary Outcome: Medical Outcome Study (MOS) Sleep Disturbance
Description: MOS Sleep Scale is a subject-rated questionnaire consisting of 12 items that assess the key constructs of sleep; assesses sleep for the 4 weeks prior to evaluation. The MOS Sleep Disturbance sub-scale scores range from 0 to 100, lower scores indicate less disturbance.
Time Frame: Week 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. MOS was measured at baseline and Week 8. For subjects not completing the study, their final data were considered Week 8 data; those without final data were excluded from analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 74
score on scale | 28.96 (1.550) [25.90 to 32.01] | 34.58 (2.237) [30.17 to 38.99]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Sleep Disturbance Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.034, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = -5.62, 95% CI [-10.82 to -0.42], Standard Error of Mean 2.639

10. Secondary Outcome: Medical Outcome Study (MOS) Snoring Score
Description: MOS Sleep Scale is a subject-rated questionnaire consisting of 12 items that assess the key constructs of sleep; assesses sleep for the 4 weeks prior to evaluation. The MOS Snoring sub-scale scores range from 0 to 100, lower scores indicate less snoring.
Time Frame: Week 8
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
score on scale | 34.21 (1.964) [30.34 to 38.08] | 29.16 (2.788) [23.66 to 34.65]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Snoring Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.128, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = 5.05, 95% CI [-1.47 to 11.58], Standard Error of Mean 3.309

11. Secondary Outcome: Medical Outcome Study (MOS) Awaken Short of Breath or Headache
Description: MOS Sleep Scale is a subject-rated questionnaire consisting of 12 items that assess the key constructs of sleep; assesses sleep for the 4 weeks prior to evaluation. The MOS Awaken Short of Breath or with a Headache sub-scale scores range from 0 to 100, lower scores indicate less difficulty.
Time Frame: Week 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. MOS was measured at baseline and Week 8. For subjects not completing the study, their final data were considered Week 8 data; those without final data were excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
score on scale | 6.90 (1.116) [4.70 to 9.09] | 9.98 (1.590) [6.85 to 13.12]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Awaken Short of Breath or Headache Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.103, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = -3.09, 95% CI [-6.81 to 0.63], Standard Error of Mean 1.887

12. Secondary Outcome: Medical Outcome Study (MOS) Sleep Quantity
Description: MOS Sleep Scale is a subject-rated questionnaire consisting of 12 items that assess the key constructs of sleep; assesses sleep for the 4 weeks prior to evaluation. The MOS Sleep Quantity sub-scale scores range from 0 to 24 (number of hours slept).
Time Frame: Week 8
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
score on scale | 6.46 (0.108) [6.25 to 6.67] | 6.02 (0.154) [5.72 to 6.33]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Sleep Quantity Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.018, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = 0.44, 95% CI [0.08 to 0.80], Standard Error of Mean 0.182

13. Secondary Outcome: Medical Outcome Study (MOS) Optimal Sleep: Number of Participants With Optimal Sleep
Description: MOS Sleep Scale is a subject-rated questionnaire consisting of 12 items that assess the key constructs of sleep; assesses sleep for the 4 weeks prior to evaluation. The MOS Optimal Sleep sub-scale score is a binary outcome derived from Sleep Quantity (SQ): the response is YES (or 1) if SQ = 7 or 8 hours per night.
Time Frame: Week 8
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
participants
  No | 85 | 44
  Yes | 73 | 31
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Optimal Sleep Optimal Sleep is a binary outcome derived from Sleep Quantity (SQ): the response is YES (or 1) if SQ = 7 or 8 hours per night. Odds ratio measured the odds of optimal sleep in pregabalin to that in placebo. "Standard Error of the Mean" equals "Standard Error of the Odds Ratio (OR)"; Test type: Superiority or Other; p = .504, Regression, Logistic — All statistical testing was 2-sided and was conducted at the 5% level of significance; OR estimated from model with Optimal sleep status (Yes/No) as response variable, and treatment, baseline Optimal sleep status as explanatory variables; Odds Ratio (OR) = 1.23, 95% CI [0.67 to 2.24], Standard Error of Mean 0.37 — The OR estimates ratio of "Odds of optimal sleep" between Pregabalin and Placebo (ie, the former to the latter). "Odds of optimal sleep" in treatment group is ratio of "Probability of having optimal sleep" vs "Probability of Not having optimal sleep"

14. Secondary Outcome: Medical Outcome Study (MOS) Sleep Adequacy
Description: MOS Sleep Scale is a subject-rated questionnaire consisting of 12 items that assess the key constructs of sleep; assesses sleep for the 4 weeks prior to evaluation. The MOS Sleep Adequacy sub-scale scores range from 0 to 100, higher scores indicate greater sleep adequacy.
Time Frame: Week 8
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 157 | 75
score on scale | 48.81 (2.244) [44.38 to 53.23] | 46.65 (3.194) [40.36 to 52.95]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Sleep Adequacy Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.571, General Linear model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = 2.15, 95% CI [-5.33 to 9.63], Standard Error of Mean 3.796

15. Secondary Outcome: Medical Outcome Study (MOS) Somnolence
Description: MOS Sleep Scale is a subject-rated questionnaire consisting of 12 items that assess the key constructs of sleep; assesses sleep for the 4 weeks prior to evaluation. The MOS Somnolence sub-scale scores range from 0 to 100, lower scores indicate less somnolence.
Time Frame: Week 8
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 74
score on scale | 34.02 (1.394) [31.28 to 36.77] | 29.31 (1.977) [25.42 to 33.21]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Somnolence Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.046, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = 4.71, 95% CI [0.08 to 9.34], Standard Error of Mean 2.349

16. Secondary Outcome: Medical Outcome Study (MOS) Overall Sleep Problems Index
Description: MOS Sleep Scale is a subject-rated questionnaire consisting of 12 items that assess the key constructs of sleep; assesses sleep for the 4 weeks prior to evaluation. The MOS Overall Sleep Problems Index is a 9-item sub-scale; scores range from 0 to 100, lower scores indicate fewer sleep problems.
Time Frame: Week 8
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 157 | 73
score on scale | 32.27 (1.204) [29.90 to 34.65] | 34.40 (1.730) [30.99 to 37.81]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Overall Sleep Problem Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.300, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = -2.12, 95% CI [-6.15 to 1.91], Standard Error of Mean 2.044

17. Secondary Outcome: Euro Quality of Life (QOL) (EQ-5D) Utility Score
Description: EQ-5D, a subject-completed questionnaire, assesses health-related QOL. QOL Health State Profile (HSP) is designed to record subject's level of current health across 5 domains (mobility, self-care, usual activities, pain/discomfort & anxiety/depression); scores are used to calculate EQ-5D Utility Score; range: -0.594 to 1.000 (from worst to best).
Time Frame: Week 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. EQ-5D was measured at baseline and Week 8. For subjects not completing the study, their final data were considered Week 8 data; those without final data were excluded from analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
score on scale | 0.651 (0.0192) [0.614 to 0.689] | 0.626 (0.0274) [0.572 to 0.680]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Endpoint Utility Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.429, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = 0.026, 95% CI [-0.038 to 0.090], Standard Error of Mean 0.0325

18. Secondary Outcome: Euro Quality of Life (EQ-5D) Visual Analog Scale (VAS)
Description: EQ-5D is a subject-completed questionnaire to assess health-related QOL (Health State Profile (HSP) & Visual Analog Scale (VAS)). The VAS is designed to rate the subject's current health state on a scale from 0 to 100 where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Week 8
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
score on scale | 61.53 (1.406) [58.76 to 64.30] | 58.03 (2.008) [54.07 to 61.99]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Endpoint VAS Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.142, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = 3.50, 95% CI [-1.18 to 8.18], Standard Error of Mean 2.375

19. Secondary Outcome: Hospital Anxiety and Depression Scale- Anxiety (HADS-A) Score
Description: HADS-A consists of 7 items that are assessed by a score of 0 = no anxiety to 3 = severe feeling of anxiety. The anxiety subscale determines a state of generalized anxiety (including anxious mood, restlessness, anxious thoughts, panic attacks). Score range = 0 to 21; higher scores indicate a greater intensity of anxiety
Time Frame: Week 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. HADS was measured at baseline and Week 8. For subjects not completing the study, their final data were considered Week 8 data; those without final data were excluded from analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
score on scale | 6.01 (0.242) [5.53 to 6.48] | 6.86 (0.345) [6.18 to 7.54]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Endpoint Anxiety Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.038, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = -0.85, 95% CI [-1.66 to -0.05], Standard Error of Mean 0.409

20. Secondary Outcome: Hospital Anxiety and Depression Scale- Depression (HADS-D) Score
Description: HADS-D consists of 7 items that are assessed by a score of 0 = no depression to 3 = severe feeling of depression. The depression subscale focuses on the state of lost interest and diminished pleasure response ("lowering of hedonic tone"). Score range = 0 to 21; higher scores indicate a greater intensity of depression
Time Frame: Week 8
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
score on scale | 7.54 (0.259) [7.03 to 8.05] | 7.73 (0.369) [7.00 to 8.46]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Endpoint Depression Score Pregabalin minus Placebo; Test type: Superiority or Other; p = 0.664, General Linear Model — All statistical testing was 2-sided and was conducted at the 5% level of significance; Estimated from general linear model with treatment and center as factors and baseline value as a covariate; Mean Difference (Final Values) = -0.19, 95% CI [-1.05 to 0.67], Standard Error of Mean 0.438

21. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: PGIC is a subject-rated instrument that measured change in subject's overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improved = minimally improved, much improved, and very much improved; Worse = minimally worse, much worse, and very much worse.
Time Frame: Week 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. PGIC was measured at Week 8. For subjects not completing the study, their final data were considered Week 8 data; those without final data were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 158 | 75
participants
  Improved | 118 | 54
  No change | 29 | 12
  Worse | 11 | 9
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Cochran-Mantel-Haenszel (CMH) test on the null hypothesis of no treatment difference in all centers. CMH test comparing Pregabalin to Placebo adjusted for center; Test type: Superiority or Other; p = 0.473, Cochran-Mantel-Haenszel — All statistical testing was 2-sided and was conducted at the 5% level of significance. p-value is from comparing Pregabalin versus Placebo; To apply CMH, each category is given a numerical score; the method of "modified rdit" used to assign numeric scores

22. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: CGIC is a clinician-rated instrument that assesses the subject's overall global improvement on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improved = minimally improved, much improved, and very much improved; Worse = minimally worse, much worse, and very much worse.
Time Frame: Week 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. CGIC was measured at Week 8. For subjects not completing the study, their final data were considered Week 8 data; those without final data were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 160 | 77
participants
  Improved | 117 | 51
  No change | 37 | 16
  Worse | 6 | 10
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.119, Cochran-Mantel-Haenszel — All statistical testing was 2-sided and was conducted at the 5% level of significance; To apply CMH, each category is given a numerical score; the method of "modified rdit" used to assign numeric scores

23. Secondary Outcome: Duration Adjusted Average Change (DAAC) of (Unadjusted) Mean Pain Score
Description: as for outcome 6
Time Frame: Weeks 1 to 8
Population: The ITT population consisted of subjects who received ≥1 dose of study medication and had contributed to the analysis of any efficacy parameter. For subjects who did not complete the study, the last 7 observations while on study medication were carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 161 | 77
score on scale | -1.24 (1.320) | -0.87 (1.488)

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/162 | 1/78
Other Adverse Events (participants affected / at risk) | 68/162 | 23/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=162) | Placebo (N=78)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=162) | Placebo (N=78)
Dizziness (Nervous system disorders) | 34 | 7
Somnolence (Nervous system disorders) | 22 | 4
Face oedema (General disorders) | 10 | 1
Oedema peripheral (General disorders) | 10 | 0
Weight increased (Investigations) | 9 | 1
Generalized oedema (General disorders) | 7 | 0
Nasopharyngitis (Infections and infestations) | 6 | 1
Constipation (Gastrointestinal disorders) | 4 | 1
Headache (Nervous system disorders) | 4 | 3
Dry mouth (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Palpitations (Cardiac disorders) | 2 | 2
Bulimia nervosa (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.